CLINICAL TRIAL: NCT05235282
Title: Effect of Oral Neuromuscular Training on Swallowing Function and Time Until Decannulation
Brief Title: Effect of Oral Neuromuscular Training on Swallowing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Hammel Neurorehabilitation Centre and University Research Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 764706
Record Dates: First submitted 2022-01-18; First posted 2022-02-11 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-04

CONDITIONS: Dysphagia
Keywords: Dysphagia
MeSH Terms: conditions — Deglutition Disorders | interventions — Deglutition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care + IQoro (Experimental): The intervention group receives usual training of swallowing function along with training 3 times each day with an IQoro oral screen
  Interventions: Device: IQoro; Other: Usual care for swallowing function
- Usual care (Active Comparator): The comparison group receives usual training of swallowing function
  Interventions: Other: Usual care for swallowing function

INTERVENTIONS:
Device: IQoro — An acrylic mouth guard with a pulling loop. The mouth guard is placed in the mouth of the patient on the outside of the teeth. The therapist pulls the loop in different directions and the patient try to close his/her mouth on the mouth guard to keep it inside the mouth.
  Arms: Usual care + IQoro
Other: Usual care for swallowing function — Cuff deflation, speaking valve, masako exercises, shaker exercises, coughing, stimulation of the oral cavity, neuromuscular electrical stimulation, postural control

SUMMARY:
In this randomized controlled trial the investigators wish to investigate the effect of an oral neuromuscular training device (called IQoro) on swallowing function and time until decannulation from a tracheostomy tube, in patients admitted for neurorehabilitation due to a severe acquired brain injury.

ELIGIBILITY:
Inclusion Criteria:

* Cuff tracheostomy tube

Exclusion Criteria:

* Not able to comply with IQoro exercises
* 3 weeks evaluation stay at the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Number of days from admission until decannulation | Number of days from baseline assessment until decannulation or right censoring at 365 days
  Time from admission until decannulation from a tracheostomy tube. For patients still admitted, decannulation is determined from the clinicians and documented i medical records. For discharged patients, decannulation is determined through medical records.

SECONDARY OUTCOMES:
Fiberoptic Endoscopic Dysphagia Severity Scale (FEDSS) | Baseline and after four weeks
  FEDSS is a scale used for Fiberoptic Endoscopic Evaluation of Swallowing. FEDSS range is 1-6, with lower scores representing better outcome
Penetration Aspiration Scale (PAS) | Baseline and after four weeks
  PAS is a scale used for Fiberoptic Endoscopic Evaluation of Swallowing. PAS range is 1-8, with lower scores representing better outcome
Yale Pharyngeal Residue Scale | Baseline and after four weeks
  Yale Pharyngeal Residue Scale is a scale used for Fiberoptic Endoscopic Evaluation of Swallowing. The Yale Scale encompass two subscales with score 1-5 on each scale, with 1 representing better outcome.
Milliliters of saliva above the cuff | Daily measures for up to four weeks
  Daily amount of saliva above the cuff of the tracheostomy tube
Functional oral intake (FOIS) | Baseline and after four weeks
  FOIS range is 1-7, with 7 representing better outcome
Iowa Oral Performance Instrument (IOPI) | Baseline and after four weeks
  Lip strength measured with the IOPI. Measured in Pascal with greater values representing greater strength

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Fabricius, PhD, Principal Investigator — Hammel Neurorehabilitation Centre and University Research Clinic
Locations (1):
- Hammel Neurorehabilitation Centre and University Research Clinic, Hammel, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No